CLINICAL TRIAL: NCT03348839
Title: Multicentre Trial, With Stepped Wedge Randomized Controled Clusters, on Medico-economic Impacts of NeLLY Service for Not on Dialysis Severe Chronic Kidney Disease
Brief Title: Medico-economic Impacts of NeLLY Service for Not on Dialysis Severe Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Calydial (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PRME-16-0418
Record Dates: First submitted 2017-11-14; First posted 2017-11-21 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-11

CONDITIONS: Chronic Kidney Disease stage4; Kidney Diseases
Keywords: telemedicine; telemonitoring; educational therapy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Multicentre study, in randomized mastered clusters, in stepped wedge
Masking Description: no one
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cluster 1 (Experimental): NeLLY service is implemented after 8 months.
  Interventions: Device: NeLLY service
- Cluster 2 (Experimental): NeLLY service is implemented after 12 months.
  Interventions: Device: NeLLY service
- Cluster 3 (Experimental): NeLLY service is implemented after 16 months.
  Interventions: Device: NeLLY service
- Cluster 4 (Experimental): NeLLY service is implemented after 20 months.
  Interventions: Device: NeLLY service
- Cluster 5 (Experimental): NeLLY service is implemented after 24 months.
  Interventions: Device: NeLLY service
- Cluster 6 (Experimental): NeLLY service is implemented after 28 months.
  Interventions: Device: NeLLY service
- Cluster 7 (Experimental): NeLLY service is implemented after 32 months.
  Interventions: Device: NeLLY service

INTERVENTIONS:
Device: NeLLY service — Telesurveillance and therapeutic support
  Other Names: Ap'Telecare

SUMMARY:
This medico-economic research project (PRME) aim to analyse NeLLY service efficiency for not on dialysis severe chronic kidney disease (DFG < 30ml/mn) patients care. NeLLY is a service that includes telemonitoring, educational therapy and support for patients with severe chronic kidney disease.

DETAILED DESCRIPTION:
NeLLY study is a multicentre trial, with stepped wedge randomized controled clusters. 2 strategies will be compared: usual patients follow-up and NeLLY service. The primary endpoint of the study is incremental cost-effectiveness ratio. This 3 years study will include 600 French patients.

NeLLY service, offering telemonitoring, educational therapy and support to patients with severe chronic kidney disease, is based on an app, both for patients and health professionals, named Ap'Telecare (@TMM).

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic kidney disease stage 4
* patient with at least 1 cardiovascular comorbidity and / or diabetes
* patient with internet connexion from home
* patient having given his express consent

Exclusion Criteria:

* dialysed patient
* refusal of patient to take part in the research
* impairment of vital prognosis within a short period
* patient expecting a transplant from a living donor within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio | Data collection all along the study: 3 years
  The primary endpoint of the study is incremental cost-effectiveness ratio comparing 2 strategies : usual patients follow-up and NeLLY service

SECONDARY OUTCOMES:
Evaluation of costs related to each strategy | Data collection every 4 months at least, all along the study: 3 years
  All medical expenses will be collected in the case report form
Evaluation of quality of life related to each strategy | every 4 months, all along the study: 3 years
  Specific questionnaire analysing patient's mobility, autonomy, pain and discomfort, anxiety and depression (patient's answer can be yes or no)
Evaluation of the financial impact of NeLLY service implementation in France | Data collection every 4 months at least, all along the study: 3 years
  All medical expenses will be collected in the case report form
Evaluation of clinical impact of NeLLY service | Data collection all along the study: 3 years
  The question is: does NeLLY reduce hospitalisation, slow chronic kidney disease evolution, increase blood pressure control. Data will be collected during usual nephrology consultations.
Evaluation of NeLLY service impacts on dialysis and transplant | Data collection all along the study: 3 years
  The question is: does NeLLY delay resorting to dialysis, avoid emergency dialysis, encourage transplant
Evaluation of NeLLY service impacts on compliance of patients | 4 times during the study: 3 years
  Specific questionnaire:
  Did the patient forget this morning to take medication? Since his last consultation, did the patient already miss any medication at home? Is the patient sometimes late to take medication? Did the patient already forget medication because of a lapse of memory? Did the patient already miss to take a medication because the patient think it can do more harm than good? Do the patient believe having too many medication to take? Patient's answer can be yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: CAILLETTE BEAUDOIN Agnès, Principal Investigator — Calydial
Locations (10):
- France (10):
  - CHU Caen, Caen
  - CHU Chalon, Chalon-sur-Saône
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Centre hospitalier Saint Joseph Saint Luc, Lyon
  - CHU Marseille, Marseille
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - ARTIC 42, Saint-Etienne
  - CHU Saint Etienne, Saint-Etienne
  - CALYDIAL, Vienne

IPD SHARING:
Plan to Share IPD: No